CLINICAL TRIAL: NCT00144209
Title: Swiss Restless Legs Syndrome Trial (SRLS) A Double-blind, Randomised, Crossover Trial Investigating the Efficacy and Safety of the Dopamine Agonist Pramipexole (Sifrol®, 0.25-0.75 mg Per Day) Versus Levodopa / Benserazide (Madopar® DR, 125-375 mg Per Day) in Patients With Restless Legs Syndrome
Brief Title: Assess Efficacy and Safety of the Dopamine Agonist Pramipexole Versus Levodopa / Benserazide (Madopar® DR) in Patients With Restless Legs Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 248.518
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pramipexole; Levodopa; Benserazide

INTERVENTIONS:
Drug: pramipexole
Drug: levodopa in combination with benserazide

SUMMARY:
The primary objective of this study is to determine that pramipexole (Sifrol) 0.25 mg to 0.75 mg daily is not inferior to levodopa 100 mg to 300 mg (in combination with benserazide 25mg to 75mg = Madopar DR) daily in the treatment of patients with idiopathic restless legs syndrome fulfilling the International Diagnostic Criteria. The efficacy parameters include an objective measure of the leg movements during the time spent in bed, and a quantitative clinical assessment of the severity of RLS, in the form of the RLS-score. In addition, the efficacy evaluations aim at comparing the impact of pramipexole and levodopa on outcome measures such as quality of life and sleep.

ELIGIBILITY:
Inclusion criteria:

* Patients diagnosed with idiopathic restless legs syndrome fulfilling the International Diagnostic Criteria 1 .
* Male or female patients, aged 25 to 85 years.
* Patients presenting RLS symptoms almost every day, as judged by the investigator and with more than 5 PLM/h during bedtime in each of three screening actigraphy nights.
* Patients must have given written informed consent in accordance with ICH-GCP and local legislation prior to participation in the study.

Exclusion criteria:

* Patients with significant diseases other than restless legs syndrome will be excluded. A significant disease is defined as a disease that, which in the opinion of the investigator may put the patient at a risk because of the participation in the study, that may influence the result of the study or the patient's ability to participate or that is expected to relevantly reduce life expectancy.
* Patients with known hypersensitivity or contraindications to pramipexole, levodopa or benserazide or any other substances present in the study medications.
* Patients with iron-deficiency
* Patients with disabilities or other incapacities that preclude regular attendance at clinic for the study visits, and patients on a shift-work-schedule or who are otherwise unable to follow a regular sleep-wake cycle.
* Patients who have been previously treated with pramipexole or levodopa.
* Pregnant or nursing women or women of childbearing age who are at risk of pregnancy and are not willing to use adequate contraceptive methods (hormonal contraception or intrauterine devices) during the study period.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-02; Primary Completion 2005-02 (Actual); Study Completion 2005-02

PRIMARY OUTCOMES:
Frequency of periodic limb movements while in bed (PLM-I) | after 4 weeks

SECONDARY OUTCOMES:
Changes in RLS-score | after 4 weeks
Changes in sleep quality as assessed in a sleep diary | after 4 weeks
Changes in Quality of Life (SF-36) | after 4 weeks
Mood changes measured by Hospital Anxiety and Depression Scale (HAD) | after 4 weeks
Overall impression assessed by Clinical Global Impression (CGI) | after 4 weeks
Changes in daytime sleepiness as assessed by the Epworth Sleepiness Scale (ESS) | after 4 weeks
Incidence and Intensity of Adverse events | up to 10 weeks
Changes in safety laboratory values | up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Schweiz GmbH.
Locations (5):
- Switzerland (5):
  - Boehringer Ingelheim Investigational Site, Bad Zurzach
  - Boehringer Ingelheim Investigational Site, Basel
  - Boehringer Ingelheim Investigational Site, Bern
  - Boehringer Ingelheim Investigational Site, Lugano
  - Boehringer Ingelheim Investigational Site, Zurich

REFERENCES:
- [Derived] Bassetti CL, Bornatico F, Fuhr P, Schwander J, Kallweit U, Mathis J; Swiss RLS study group. Pramipexole versus dual release levodopa in restless legs syndrome: a double blind, randomised, cross-over trial. Swiss Med Wkly. 2011 Nov 21;141:w13274. doi: 10.4414/smw.2011.13274. eCollection 2011. PMID 22101745
- [Derived] Kallweit U, Khatami R, Pizza F, Mathis J, Bassetti CL. Dopaminergic treatment in idiopathic restless legs syndrome: effects on subjective sleepiness. Clin Neuropharmacol. 2010 Nov-Dec;33(6):276-8. doi: 10.1097/WNF.0b013e3181fd82a1. PMID 21060282